CLINICAL TRIAL: NCT00417534
Title: Genetic Predisposition of Coronary Artery Disease in Patients Verified With Coronary Angiogram The COROGENE-Study
Brief Title: Genetic Predisposition of Coronary Artery Disease -- The COROGENE-Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Helsinki (Other)
Other Study IDs: 214841
Record Dates: First submitted 2006-12-29; First posted 2007-01-01 (Estimated); Last update posted 2007-07-03 (Estimated); Status verified 2006-12

CONDITIONS: Coronary Disease; Inflammation
Keywords: Coronary Disease; Inflammation; Genetics; HLA Antigens; Aortic Valve
MeSH Terms: conditions — Coronary Disease; Inflammation

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
The aim of this study is to identify genetic loci,or gene variations contributing to inflammation and to the development of CHD. We will compare coronary angiogram results to genetic findings within coronary artery disease patients and in patients with normal coronaries.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is a chronic inflammatory disease, progression of which may be accelerated by immunological mechanisms. Genes involved in regulation of inflammation and protection against infectious agents may affect picture of the disease . Major Histocompatibility Complex (MHC) region carries genes involved in innate and adaptive immunity and inflammation. We have for the first time, identified genetic factors located in HLA region, showing several fold risk for disease predisposition likely forming an important component to explain the high incidence of coronary heart disease in the Finnish population.

The aim of this study is to rerun our preliminary results, and further identify genetic loci, or gene variations contributing to the development of CHD. The strategy is to collect altogether 5000 patients assigned to coronary angiogram in Helsinki University Central Hospital. We will compare the angiogram results to genetic findings first in patients with normal coronaries, and in patients with different stages of CHD. Secondly we will compare phenotypic changes in inflammation and try to find out if the phenotype differs in different genotypes. Thirdly we will collect patients from hospital discharge registry, and compare mortality and morbidity results in different gene groups.

Finally, we aim to record echocardiograms of the aortic valves in altogether 3500 consecutive patients undergoing coronary angiography. We try to identify genetic loci and gene variations contributing to the fibrosis and calcification of the aortic valve.

The results of the study provide a possibility to develop a gene test to recognize patients at risk at its early stage, and needing for preventive medicine.

ELIGIBILITY:
Inclusion Criteria:

* Patient assigned to coronary angiogram

Exclusion Criteria:

* Inability to give informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2006-06; Study Completion 2009-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Juha P Sinisalo, MD, PhD, Principal Investigator — Helsinki University Central Hospital, Division of Cardiology
Locations (1):
- Helsinki University Central Hospital, Division of Cardiology, Helsinki, Finland

REFERENCES:
- [Background] Hansson GK. Inflammation, atherosclerosis, and coronary artery disease. N Engl J Med. 2005 Apr 21;352(16):1685-95. doi: 10.1056/NEJMra043430. No abstract available. PMID 15843671
- [Background] Sinisalo J, Mattila K, Valtonen V, Anttonen O, Juvonen J, Melin J, Vuorinen-Markkola H, Nieminen MS; Clarithromycin in Acute Coronary Syndrome Patients in Finland (CLARIFY) Study Group. Effect of 3 months of antimicrobial treatment with clarithromycin in acute non-q-wave coronary syndrome. Circulation. 2002 Apr 2;105(13):1555-60. doi: 10.1161/01.cir.0000012544.07696.1f. PMID 11927522
- [Background] Ye Z, Liu EH, Higgins JP, Keavney BD, Lowe GD, Collins R, Danesh J. Seven haemostatic gene polymorphisms in coronary disease: meta-analysis of 66,155 cases and 91,307 controls. Lancet. 2006 Feb 25;367(9511):651-8. doi: 10.1016/S0140-6736(06)68263-9. PMID 16503463
- [Background] Swanberg M, Lidman O, Padyukov L, Eriksson P, Akesson E, Jagodic M, Lobell A, Khademi M, Borjesson O, Lindgren CM, Lundman P, Brookes AJ, Kere J, Luthman H, Alfredsson L, Hillert J, Klareskog L, Hamsten A, Piehl F, Olsson T. MHC2TA is associated with differential MHC molecule expression and susceptibility to rheumatoid arthritis, multiple sclerosis and myocardial infarction. Nat Genet. 2005 May;37(5):486-94. doi: 10.1038/ng1544. Epub 2005 Apr 10. PMID 15821736
- [Background] Saikku P, Leinonen M, Mattila K, Ekman MR, Nieminen MS, Makela PH, Huttunen JK, Valtonen V. Serological evidence of an association of a novel Chlamydia, TWAR, with chronic coronary heart disease and acute myocardial infarction. Lancet. 1988 Oct 29;2(8618):983-6. doi: 10.1016/s0140-6736(88)90741-6. PMID 2902492
- [Background] Lusis AJ, Mar R, Pajukanta P. Genetics of atherosclerosis. Annu Rev Genomics Hum Genet. 2004;5:189-218. doi: 10.1146/annurev.genom.5.061903.175930. PMID 15485348
- [Background] Paavonen KJ, Chapman H, Laitinen PJ, Fodstad H, Piippo K, Swan H, Toivonen L, Viitasalo M, Kontula K, Pasternack M. Functional characterization of the common amino acid 897 polymorphism of the cardiac potassium channel KCNH2 (HERG). Cardiovasc Res. 2003 Sep 1;59(3):603-11. doi: 10.1016/s0008-6363(03)00458-9. PMID 14499861
- [Background] Ozaki K, Ohnishi Y, Iida A, Sekine A, Yamada R, Tsunoda T, Sato H, Sato H, Hori M, Nakamura Y, Tanaka T. Functional SNPs in the lymphotoxin-alpha gene that are associated with susceptibility to myocardial infarction. Nat Genet. 2002 Dec;32(4):650-4. doi: 10.1038/ng1047. Epub 2002 Nov 11. PMID 12426569
- [Derived] Sinisalo J, Vlachopoulou E, Marchesani M, Nokelainen J, Mayranpaa MI, Lappalainen J, Paakkanen R, Wennerstrom A, Salli K, Niemi HJ, Mannisto S, Salo P, Junttila J, Eskola M, Nikus K, Arstila TP, Perola M, Huikuri H, Karhunen PJ, Kovanen PT, Palotie A, Havulinna AS, Lluis-Ganella C, Marrugat J, Elosua R, Salomaa V, Nieminen MS, Lokki ML. Novel 6p21.3 Risk Haplotype Predisposes to Acute Coronary Syndrome. Circ Cardiovasc Genet. 2016 Feb;9(1):55-63. doi: 10.1161/CIRCGENETICS.115.001226. Epub 2015 Dec 17. PMID 26679868